CLINICAL TRIAL: NCT03592784
Title: Carbohydrate-Last Food Order Intervention for Gestational Diabetes Mellitus
Brief Title: Food Order Intervention for Gestational Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment during Covid pandemic, however sufficient data gathered for assessment of primary outcome
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1802018956
Record Dates: First submitted 2018-06-18; First posted 2018-07-19 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Nutrition Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food Order Therapy + Medical Nutrition Therapy (Experimental)
  Interventions: Behavioral: Food Order Therapy; Behavioral: Medical Nutrition Therapy
- Medical Nutrition Therapy Alone (Active Comparator)
  Interventions: Behavioral: Medical Nutrition Therapy

INTERVENTIONS:
Behavioral: Food Order Therapy — Instructing patient to, whenever possible, eat carbohydrates at the end of their meal.
  Arms: Food Order Therapy + Medical Nutrition Therapy
Behavioral: Medical Nutrition Therapy — Key components of this therapy include counseling to incorporate portion control, increased intake of vegetables and low glycemic index carbohydrates, and mild carbohydrate restriction.

SUMMARY:
This is a randomized controlled feasibility trial for women diagnosed with gestational diabetes mellitus (GDM). The current front-line treatment for GDM is medical nutrition therapy (MNT), i.e. personalized diets which may or may not include mild carbohydrate restriction. Use of carbohydrate restriction increases the risk of the mother developing ketosis, a harmful condition for both the mother and fetus. If MNT is not enough to stabilize blood sugar levels, then pharmaceuticals are prescribed. In patients with type-2 diabetes and prediabetes, the carbohydrate-last food order behavior has been shown to improve post-meal blood sugar control without the need of reduced carbohydrate intake. Given this data, the addition of this intervention to MNT in patients with GDM may be helpful in achieving controlled blood sugar levels without increasing the risk of ketosis. This study will include two randomized groups diagnosed with GDM. Patients in the control group will be prescribed standard MNT. Patients in the intervention group will have identical MNT but with additional food order instruction/therapy. All patients will be followed up with at 1-2 week intervals. At each follow-up the physician and dietician will analyze the patient's blood sugar measurements and, among additional factors, determine if pharmaceuticals should be added. Treatment will continue through delivery. The primary aim of this study is to assess the feasibility of the carbohydrate last food order in GDM and generate preliminary data on its effects on glucose control.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant subjects ≥18 years old
* Newly diagnosed with GDM between 24-32 weeks of gestation with at least 2 days of self-monitored glucose logs or diagnosed via a 50g glucose challenge test (GCT) greater than 200mg/dL

Exclusion Criteria:

* Pre-existing diabetes prior to conception
* Patients whom do not plan on consuming at least 3 meals daily throughout gestation (e.g. during Ramadan)
* Requirement of special medical diet (e.g. from phenylketonuria, celiac disease, etc.)
* History of bariatric surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-04-22 (Actual)

PRIMARY OUTCOMES:
Feasibility of the Food Order Intervention | 8 weeks
  Measured via feasibility questionnaire.

SECONDARY OUTCOMES:
Average 1-hour postprandial glucose | 2, 4, 6, 8, 10, 12 weeks
  Averaged from self-monitored blood glucose logs.
Time to initiation of pharmacotherapy | 2, 4, 6, 8, 10, 12 weeks
  Measured in weeks from enrollment in the study.
Proportion of patients requiring the addition of pharmacotherapy | Week 16 or End of study (at delivery)
  Measured as a percentage of patients in each arm.
Birthweight | Week 16 or End of study (delivery)
  Measured in lbs.

CONTACTS AND LOCATIONS:
Overall Officials: Alpana P Shukla, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Materal-Fetal Medicine of Weill Cornell Medicine, New York, New York, United States